CLINICAL TRIAL: NCT07235943
Title: Therapeutic Low Laser Therapy and Kinesio Taping in Patients With Grade 1 and Grade 2 Lateral Ankle Sprain
Brief Title: Therapeutic Low Laser Therapy and Kinesio Taping for Lateral Ankle Sprain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lahore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: UOL/IREB/25/09/0059
Record Dates: First submitted 2025-08-26; First posted 2025-11-19 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2024-09

CONDITIONS: Lateral Ankle Sprain; Ankle Sprain 1St Degree; Ankle Sprain 2Nd Degree
Keywords: Low-Level Laser Therapy (LLLT); Kinesio Taping; Ankle Injury Rehabilitation; Lateral Ankle Sprain; Grade 1 Ankle Sprain; Grade 2 Ankle Sprain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental)
  Interventions: Other: Combined: Low Laser Therapy with Kinesio Taping
- Group B (Active Comparator)
  Interventions: Other: Using Low-Level Laser Therapy

INTERVENTIONS:
Other: Using Low-Level Laser Therapy — 1. Initial Assessment:
     Comprehensive evaluation is necessary to ascertain the degree of ankle sprain (Grade 1 or Grade 2), range of motion, discomfort, swelling, and functional restrictions at the beginning of treatment.
     * Grade 1 Sprain: Minimal swelling, mild ligament stretching, and no significant impairment of function.
     * Grade 2 Sprain: Moderate swelling, pain while bearing weight, reduced range of motion, and partial ligament treatment
  2. Low-Level Laser Therapy (LLLT) Treatment
     * General Principles of LLLT for Ankle Sprains Purpose: LLLT is used to improve circulation, lessen pain and inflammation, and promote tissue repair.
  Mechanism of Action: By promoting mitochondrial activity, LLLT raises the synthesis of collagen and ATP. By releasing endorphins and increasing nitric oxide, it improves circulation, lowers inflammation, and regulates pain.
  LLLT parameters for lateral ankle sprains in grades 1 and 2
  • Wavelength: For deeper tissue penetration (targeting ligaments and te
  Arms: Group B
Other: Combined: Low Laser Therapy with Kinesio Taping — Low-Level Laser Therapy (LLLT) Treatment
  * General Principles of LLLT for Ankle Sprains
  * Purpose: LLLT is used to improve circulation, lessen pain and inflammation, and promote tissue repair.
  * Mechanism of Action: By promoting mitochondrial activity, LLLT raises the synthesis of collagen and ATP. By releasing endorphins and increasing nitric oxide, it improves circulation, lowers inflammation, and regulates pain.
    2. LLLT parameters for lateral ankle sprains in grades 1 and 2 (initial step)
  * Wavelength: For deeper tissue penetration (targeting
    2. Kinesio Taping Application (Second Step) Kinesio taping is performed to support and stabilize the area of injury. By reducing discomfort and swelling, it may enhance comfort during activities.
  For Grade 1 Sprains (Mild Injury) Technique:
  1. Y-Strip for Lateral Ankle Sprain: Place the tape at the base of the fifth metatarsal, or the dorsum of the foot.
  2. Wrap Around the Lateral Ankle: Wrap the two Y-shape tails around the lateral ankle,
  Arms: Group A

SUMMARY:
HYPOTHESIS

Null Hypothesis (H0):

There is no significant effect of therapeutic low laser therapy and kinesio taping in patients with grade 1 & 2 lateral ankle sprain.

Alternative Hypothesis (HA):

There is a significant effect of therapeutic low laser therapy and kinesio taping in patients with grade 1 & 2 lateral ankle sprain.

ELIGIBILITY:
Inclusion Criteria:

* Participants are of both genders
* Patients age will be from 20-40 years
* Sub-acute ankle sprains (<2 weeks post-injury)
* Grade 1& 2 lateral ankle sprains
* A clinical diagnosis of at least one prior severe ankle sprain is required
* Sensations of the ankle joint that it may "give way", recurrent sprain, or "looseness"
* A score of Identification of Functional Ankle Instability of at least 11 (if both sides are equal, the lower functional side will be chosen)
* Not allergic to KT

Exclusion Criteria:

* Patients with a history of prior injury to the back, hip, knee, or severe injury to the ankle in the last two years
* Systemic diseases like Rheumatoid arthritis, Diabetics, Neuropathies
* Ankle fracture, subluxation, dislocation
* The patient has received an intra-articular steroid injection in any recent operation of either of the two lower limbs.
* Psychological disorders
* Any spinal surgery

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 62 (Actual)
Dates: Start 2024-11-24 (Actual); Primary Completion 2025-03-22 (Actual); Study Completion 2025-05-30 (Actual)

PRIMARY OUTCOMES:
Foot and Ankle Disability Index | Baseline and at 12 weeks
  The 34-item Foot and Ankle Disability Index is broken down into two subscales: the Foot and Ankle Disability Index and the Foot and Ankle Disability Index Sport. FADI has 26 items, whereas FADI Sport has only 8 items. FADI consists of 4 items dealing with pain and 22 items dealing with activities. 8 items in FADI-Sport are activity related. It tests more complex aspects that are crucial to sports. In contrast to FADI, FADI Sport is a subscale derived from the original population scale and specifically tailored for athletes. It is designed to fill this need by identifying the lower-functioning subjects in terms of the higher functions
Numeric Pain Rating Scale (NPRS) | Baseline and at 12 weeks
  An outcome measure that provides a unidimensional gauge of pain intensity in adults. A respondent chooses an integer between 0 (no pain) and 10 (worst possible pain). Higher scores indicate greater pain severity.
RANGE OF MOTION | Baseline and at 12 weeks
  Range of Motion is the maximum movement a joint can achieve, assessed through active (AROM) and passive (PROM) methods, typically measured in degrees using a goniometer. Higher values indicate greater mobility.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Lahore, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kobayashi T, Suzuki D, Kondo Y, Tokita R, Katayose M, Matsumura H, Fujimiya M. Morphological characteristics of the lateral ankle ligament complex. Surg Radiol Anat. 2020 Oct;42(10):1153-1159. doi: 10.1007/s00276-020-02461-3. Epub 2020 Mar 30. PMID 32227271
- [Background] Ghozy S, Dung NM, Morra ME, Morsy S, Elsayed GG, Tran L, Minh LHN, Abbas AS, Loc TTH, Hieu TH, Dung TC, Huy NT. Efficacy of kinesio taping in treatment of shoulder pain and disability: a systematic review and meta-analysis of randomised controlled trials. Physiotherapy. 2020 Jun;107:176-188. doi: 10.1016/j.physio.2019.12.001. Epub 2019 Dec 9. PMID 32026818
- [Background] Gaddi D, Mosca A, Piatti M, Munegato D, Catalano M, Di Lorenzo G, Turati M, Zanchi N, Piscitelli D, Chui K, Zatti G, Bigoni M. Acute Ankle Sprain Management: An Umbrella Review of Systematic Reviews. Front Med (Lausanne). 2022 Jul 7;9:868474. doi: 10.3389/fmed.2022.868474. eCollection 2022. PMID 35872766
- [Background] Abdelbasset WK, Nambi G, Alsubaie SF, Abodonya AM, Saleh AK, Ataalla NN, Ibrahim AA, Tantawy SA, Kamel DM, Verma A, Moawd SA. A Randomized Comparative Study between High-Intensity and Low-Level Laser Therapy in the Treatment of Chronic Nonspecific Low Back Pain. Evid Based Complement Alternat Med. 2020 Oct 28;2020:1350281. doi: 10.1155/2020/1350281. eCollection 2020. PMID 33178306